CLINICAL TRIAL: NCT04404140
Title: A Phase Ib, Open-Label, Multicenter Study Evaluating The Safety, Efficacy and Pharmacokinetics Of Ipatasertib In Combination With Atezolizumab And Docetaxel In Metastatic Castration-Resistant Prostate Cancer.
Brief Title: A Study Evaluating The Safety, Efficacy and Pharmacokinetics Of Ipatasertib In Combination With Atezolizumab And Docetaxel In Metastatic Castration-Resistant Prostate Cancer (mCRPC).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Despite many risk-minimization strategies, the combination of ipatasertib, atezolizumab and docetaxel was challenging due to multiple study treatment modifications required to manage toxicity, making further enrollment inappropriate.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO41792; 2019-004591-19 (EudraCT Number)
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Castration-Resistant Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — ipatasertib; atezolizumab; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipatasertib + Atezolizumab + Docetaxel (Experimental): Part A (Safety Run-In): 12 Participants will be administered Ipatasertib orally once a day [QD] from Day 1 to Day 14 in combination with Atezolizumab administered by intravenous (IV infusion) every 3 weeks (Q3W) on Day 1 of each cycle (a cycle being 21 days) and Docetaxel administered by IV infusion (Q3W) on Day 1 of each cycle. Docetaxel will be administered for a maximum of 10 cycles (approximately 7 months), after which Atezolizumab and Ipatasertib will be administered as a doublet until disease progression. During Part A, a staggered recruitment will be applied to the first and potentially first 6 participants to enrol a participant only once the former one has safely overcome the safety time window (Cycle 1).
  Part B (Expansion): 38 Participants will be administered Ipatasertib, Atezolizumab and Docetaxel as described above, though without a staggered enrolment or safety assessment window.
  Interventions: Drug: Ipatasertib; Drug: Atezolizumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered at a dose of 400 mg, as per the dosing schedule described above.
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose of 1200 mg, as per the dosing schedule described above.
Drug: Docetaxel — Docetaxel will be administered at a dose of 75 mg/m^2, as per the dosing schedule described above.

SUMMARY:
A study evaluating the safety, preliminary efficacy and pharmacokinetics of ipatasertib in combination with atezolizumab and docetaxel in participants with mCRPC previously treated with second-generation AR (Androgen Receptor)-targeted therapy. The study consists of two parts: [1] Part A: Safety run-in cohort of approximately 12 participants; [2] Part B: Expansion cohort of approximately 38 participants. All participants in this study will continue to be treated until progression of disease, loss of clinical benefit, unacceptable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol.
* Adenocarcinoma of the prostate without small-cell or neuroendocrine features.
* Metastatic disease that cannot be treated with curative intent.
* Surgical or medical castration with testosterone serum level < 50 ng/dL (1.7 nM).
* For participants treated with luteinizing hormone-releasing hormone analogs, initiation therapy >= 4 weeks prior to the first dose of study treatment and continued therapy throughout study treatment.
* Progression of Prostate Cancer.
* Receipt of at least one prior line of second generation AR-targeted therapy.
* For participants in Part A of study: measurable visceral disease or measurable extrapelvic adenopathy per RECIST v1.1.
* For participants in Part B of study: either measurable visceral disease or measurable extrapelvic adenopathy by RECIST v1.1 or bone lesions by bone scan, or both.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy of >= 3 months.
* Ability to swallow oral study drug.
* Adequate organ and bone marrow function.
* Resolved or stabilized toxicities resulting from previous therapy to Grade 1 (except for alopecia and neuropathy).
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm.

Exclusion Criteria:

* Prior treatment with an AKT, PI3K, or mTOR inhibitor.
* Prior treatment with radium or other therapeutic radiopharmaceuticals for prostate cancer.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
* Prior treatment with docetaxel or another chemotherapy agent for mCRPC.
* Treatment with investigational therapy within 14 days prior to initiation of study drug.
* History or known presence of central nervous system metastases including leptomeningeal carcinomatosis.
* Uncontrolled tumor-related pain.
* Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment.
* Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco- regional therapy if appropriate prior to enrollment.
* Non-study-related minor surgical procedures =< 5 days or major (invasive) surgical procedure =< 28 days prior to the first dose of study treatment.
* Active Hepatitis B and C infection (HBV/HCV).
* Known HIV infection.
* Uncontrolled pleural effusion, pericardial effusion, or ascites.
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment.
* Malabsorption syndrome or other condition that would interfere with enteral absorption.
* Serious infection requiring antibiotics within 14 days prior to the first dose of study treatment.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study.
* History of another malignancy within 5 years prior to enrollment.
* History of clinically significant cardiovascular dysfunction.
* Presence of any other condition, metabolic dysfunction, physical examination finding, or laboratory finding that may increase the risk associated with study participation or may interfere with the interpretation of study results and in the opinion of the investigator, would make the participant inappropriate for study entry.

Ipatasertib-Specific Exclusion Criteria:

* Type 1 or Type 2 diabetes mellitus requiring insulin at study entry.
* History of inflammatory bowel disease (e.g., Crohn disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis).
* Grade >= 2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia.
* Treatment with strong CYP3A inhibitor or strong CYP3A inducer within 2 weeks or 5 drug-elimination half-lives of this treatment (whichever is longer) prior to initiation of study drug.

Atezolizumab-Specific Exclusion Criteria:

* Active or history of autoimmune disease or immune deficiency.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Prior allogeneic stem cell or solid organ transplantation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment with atezolizumab or within 5 months after the last dose of atezolizumab.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies.
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives of the drug (whichever is longer) prior to initiation of study treatment.
* Need for chronic corticosteroid therapy of >10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease.
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study.

Docetaxel-Specific Exclusion Criteria:

* Known hypersensitivity or contraindication to any component of docetaxel, including its excipient polysorbate 80.
* Grade >= 2 peripheral neuropathy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 35 months
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Confirmed Prostate Specific Antigen (PSA) Response | Up to 35 months
  Defined as the proportion of participants with a reduction in their PSA levels of 50% or more from baseline, confirmed by a second evaluation at least 3 weeks later
Overall Response Rate (ORR) (In participants presenting with measurable visceral disease or measurable extrapelvic adenopathy at baseline) | Up to 35 months
  Defined as the proportion of participants with a complete response (CR) or partial response (PR) on two consecutive occasions >= 4 weeks apart, as determined by the Investigator according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors, Version 1.1)

SECONDARY OUTCOMES:
Time to PSA Progression | Up to 35 months
radiographic Progression-Free Survival (rPFS) | Up to 35 months
  Assessed according to the Prostate Cancer Working Group 3 (PCWG3) criteria
Overall Survival (OS) (median OS and landmark survival at 12, 18 and 24 months) | Up to 35 months
Documented Objective Response (DOR) (In participants presenting with measurable visceral disease or measurable extrapelvic adenopathy at baseline) | Up to 35 months
  Defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Clinical Benefit Rate (CBR) (In participants presenting with measurable visceral disease or measurable extrapelvic adenopathy at baseline) | Up to 35 months
  Defined as the proportion of participants who have an objective response (a CR or a PR) or stable disease for at least 27 weeks, as determined by the Investigator according to RECIST v1.1 and PCWG3 criteria
Plasma Concentrations (ng/mL) of Ipatasertib and G-037720 at pre-specified timepoints | Up to 35 months
Serum Concentrations (ng/mL) of Atezolizumab at pre-specified timepoints | Up to 35 months
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Atezolizumab | Up to 35 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- France (4):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Centre Val Aurelle Paul Lamarque; Radiotherapie, Montpellier
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Gustave Roussy, Villejuif
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- Spain (2):
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
- Switzerland (2):
  - Kantonsspital Graubünden Medizin Onkologie; Onkologie und Hämatologie, Chur
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich